CLINICAL TRIAL: NCT03469050
Title: Rifaximin Delayed Release (400 mg Tablet) for the Prevention of Recurrent Acute Diverticulitis and Diverticular Complications. A Phase II, Multicenter, Double-blind, Placebo-controlled, Randomized Clinical Trial
Brief Title: Rifaximin Delayed Release for the Prevention of Recurrent Acute Diverticulitis and Diverticular Complications.
Acronym: ROAD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REDIV/002/17; 2017-002708-28 (EudraCT Number)
Record Dates: First submitted 2018-03-06; First posted 2018-03-19 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-07

CONDITIONS: Diverticulitis
Keywords: Recurrent acute diverticulitis; Prevention; Diverticular complications; Rifaximin delayed release; Diverticulitis; SIBO
MeSH Terms: conditions — Diverticulitis | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: This study is a phase II, multicenter, double-blind, placebo-controlled, randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rifaximin delayed released 800 mg b.i.d. (Experimental): (i.e. 2 x 400 mg tablet twice a day; total daily dose: 1600 mg) for 10 consecutive days a month, for 12 months
  Interventions: Drug: Rifaximin delayed released 400mg Tablet
- Rifaximin delayed released 400 mg b.i.d (Experimental): (i.e. 1x400 mg tablet plus 1 placebo tablet twice a day; total daily dose: 800 mg) for 10 consecutive days a month, for 12 months
  Interventions: Drug: Rifaximin delayed released 400mg Tablet; Other: Placebo
- Placebo b.i.d. (Placebo Comparator): (i.e. 2 x placebo tablets twice a day) for 10 consecutive days a month, for 12 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rifaximin delayed released 400mg Tablet — Rifaximin delayed released
  Other Names: Rifaximin-EIR
  Arms: Rifaximin delayed released 400 mg b.i.d; Rifaximin delayed released 800 mg b.i.d.
Other: Placebo — Placebo BID + Placebo BID
  Arms: Placebo b.i.d.; Rifaximin delayed released 400 mg b.i.d

SUMMARY:
Colonic microbiota changes may play a key role in the pathogenesis of acute diverticulitis. A previous proof-of-concept study suggests that rifaximin, a low-absorbable oral antibiotic, may be beneficial for prevention of acute diverticulitis recurrence by modulating the gut microflora.

The main objective of this study is to evaluate the safety and efficacy of two different doses of a delayed release formulation of rifaximin, versus placebo, for the prevention of recurrence of acute diverticulitis and diverticular complications in patients with a recent episode of acute diverticulitis.

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women aged 18-80 years at screening.
* Female participants must be either of non-childbearing potential or of childbearing potential with a negative pregnancy test result at screening and randomization AND agreeing to use a highly effective method of contraception.
* A previous documented episode of diverticulitis between 30 and 180 days prior to screening.
* Clinical remission from acute diverticulitis at screening

Key Exclusion Criteria:

* History of two or more acute diverticulitis episodes or history of any diverticular complication.
* Any documented current organic disease of the gastrointestinal tract other than diverticulosis
* Laboratory signs of clinically significant acute inflammation or signs/symptoms of diverticular complications.
* Diagnosis or history of inflammatory bowel disease (or other conditions associated with ulcerative lesions of the intestinal tract).
* Patients with positive Clostridium difficile toxin stool assay.
* Use of marketed rifaximin (or neomycin or other low-absorbable oral antibiotics) during or after the previous episode of acute diverticulitis.
* Severe hepatic impairment
* Severe kidney impairment
* Any other current significant health condition that in the Investigator's judgement may: i) jeopardize the patient's safe participation in the trial or ii) make unlikely the patient's completion of the study or iii) make unlikely the patient's compliance with the study procedures.
* History of hypersensitivity to rifaximin, rifamycin-derivatives or any of the rifaximin delayed release or placebo excipients.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Rate of patients with recurrence of diverticulitis and/or diverticular complications over the 12-month treatment period. | 12-month treatment period

SECONDARY OUTCOMES:
Rate of patients with an acute episode of prolonged (≥24 hours) left-lower quadrant abdominal pain plus leukocytosis/elevation of CRP [Time Frame: 12-month treatment period] | 12-month treatment period
Time to diverticulitis recurrence or complication | 12-month treatment period
Rate of patients with diverticulitis-associated fever | 12-month treatment period
Left-lower quadrant abdominal pain intensity | 12-month treatment period
Left-lower quadrant abdominal pain duration | 12-month treatment period
Number of days in a year with left-lower quadrant abdominal pain | 12-month treatment period
Number of weeks in a year with episodes of prolonged (≥24 hours) left-lower quadrant abdominal pain | 12-month treatment period
Number of days in a year with any abdominal pain | 12-month treatment period
Number of weeks in a year with bloating | 12-month treatment period
Change in bowel habits | 12-month treatment period
  Evaluated by Bristol Stool Scale
Rate of any hospitalization for diverticulitis | 12-month treatment period
Rate of hospitalization for diverticulitis without surgery | 12-month treatment period
Rate of elective surgery for diverticulitis | 12-month treatment period
Rate of emergency surgery for diverticulitis | 12-month treatment period
Change in Quality of Life | 12-month treatment period
  Evaluated by SF36 Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Blè, MD, Study Director — Alfasigma S.p.A.
Locations (64):
- France (7):
  - Hôpital Avicenne Service Gastro-entérologie, Bobigny
  - Cabinet Médical, Lille
  - Centre Hospitalier Regional Universitaire Claude Huriez Service de Chirurgie Digestive et Générale, Lille
  - Hôpital Saint-Joseph Service Hépato-Gastroentérologie, Marseille
  - CHU Nantes, Hôtel Dieu Clinique de Chirurgie digestive et endocrinienne (CCDE) Institut des maladies de l'Appareil Digestif (IMAD), Nantes
  - Hôpital Charles Nicolle - CHU Rouen Service Hépato-Gastroentérologie, Rouen
  - Centre Hospitalier Universitaire (CHU) de Strasbourg Service de Chirurgie Digestive et Endocrinienne, Strasbourg
- Germany (5):
  - Gemeinschaftspraxis - Praxis Überruhr, Essen
  - Medamed GmbH Studienambulanz Leipzig, Leipzig
  - MVZ Dres. Eisenbach, Simon, Schwarz, Leverkusen
  - Gemeinschaftspraxis Dres. Balck, Meine
  - Praxis Dres. med. Naudts und Nowack, Rodgau
- Italy (38):
  - Ospedale Cardinal Massaia SOC Gastroenterologia ed Endoscopia Digestiva, Asti
  - Ospedale Civile S. Agostino Estense - Divisione di Endoscopia Digestiva, Baggiovara
  - Azienda Ospedaliera Policlinico Consorziale di Bari Dipartimento di Gastroenterologia, Bari
  - Ospedale "San Paolo" - Unità Operativa Complessa di Gastroenterologia ed Endoscopia Digestiva, Bari
  - Università degli Studi di Bari Policlinico Medicina Interna, Bari
  - AOU di Bologna - Policlinico S.Orsola Malpighi - Dipartimento di Scienze Mediche e Chirurgiche, Bologna
  - AOU Cagliari - Policlinico Monserrato Gastroenterologia, Cagliari
  - Azienda Ospedaliera Garibaldi Unità Operativa Complessa di Gastroenterologia, Catania
  - Ospedale Ciaccio - De Lellis Divisione di Gastroenterologia ed Endoscopia Digestiva, Catanzaro
  - Policlinico Ss Annunziata - ASL 2 Lanciano Vasto Chieti UOSD Endoscopia Digestiva, Chieti
  - Ospedale Valduce Unità Operativa Complessa di Gastroenterologia, Como
  - Ospedale S. Salvatore di L'Aquila Unità Operativa di Gastroenterologia, Epatologia e Nutrizione, Coppito
  - Ospedale Civile San Giovanni di Dio - Divisione di Gastroenterologia ed Endoscopia Digestiva, Crotone
  - Ente Ospedaliero Ospedali Galliera Chirurgia Generale, Genova
  - Ospedale Policlinico S.Martino Istituto di Ricovero e Cura per l'Oncologia Dipartimento di Medicina Interna e Specialità Mediche U.O. Clinica Gastroenterologica, Genova
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - UNIMI - San Paolo (ASST Santi Paolo e Carlo) Medicina Generale, Milan
  - Ospedale San Gerardo Endoscopia Digestiva, Monza
  - AOU Seconda Università degli Studi di Napoli Unità Operativa Complessa di Epato-Gastroenterologia, Napoli
  - Policlinico Federico II - UO di Epatogastroenterologia ed endoscopia digestiva, Napoli
  - Policlinico Federico II - UOSD Diagnosi Fisiopatologica e Terapia delle Malattie Motorie Digestive, Napoli
  - AOU di Padova Unità Operativa Complessa di Gastroenterologia, Padua
  - Ospedale Buccheri La Ferla Fetebenefratelli Unità Operativa di Gastroenterologia e Endoscopia Digestiva, Palermo
  - Fondazione IRCCS Policlinico San Matteo Dipartimento di Medicina Interna, Pavia
  - PO Cisanello - AOU Pisana Unità Operativa Complessa di Gastroenterologia - AOUP Gastroenterologia Universitaria, Pisa
  - Ospedale Popoli Unità Operativa Semplice Dipartimentale Chirurgia Endoscopica, Popoli
  - Azienda Ospedaliera San Giovanni Addolorata Gastroenterologia ed Endoscopia Digestiva, Roma
  - Fondazione Policlinico Universitario A. Gemelli Unità Operativa Complessa di Gastroenterologia e Malattie del Fegato, Roma
  - Ospedale Cristo Re - Divisione di Medicina Interna e Gastroenterologia, Roma
  - Ospedale Sant'Andrea - Gastroenterologia, Roma
  - Policlinico Universitario Campus Biomedico Unità Operativa Complessa di Gastroenterologia ed Endoscopia Digestiva, Roma
  - Istituto Clinico Humanitas-Unità Operativa Malattie Infiammatorie Croniche Intestinali, Rozzano
  - AOU OO. RR. San Giovanni di Dio e Ruggi d'Aragona - Dipartimento di Medicina e Chirurgia - Gastroenterologia, Salerno
  - IRCCS Policlinico San Donato Unità Operativa Medicina Generale III, Gastroenterologia, San Donato Milanese
  - Ospedale Sant'Anna Unità Operativa di Medicina Interna, San Fermo della Battaglia
  - Azienda Ospedaliera San Giovanni Battista Molinette - S.C. Gastroenterologia e Epatologia, Torino
  - Ospedale di Circolo e Fondazione Macchi Endoscopia, Varese
  - Azienda Ospedaliera Universitaria Integrata - UOC Gastroenterologia A- Borgo Trento-Dipartimento Medicina Generale, Verona
- Netherlands (3):
  - Meander Medisch Centrum Surgery, Amersfoort
  - VU Medisch Centrum Gastroenterology, Amsterdam
  - Ikazia ziekenhuis Gastroenterology, Rotterdam
- Spain (10):
  - Hospital General Universitario de Alicante Servicio de Aparato Digestivo, Alicante
  - Centre Médic Teknon Servicio de Aparato Digestivo, Barcelona
  - Hospital Clínic Servicio de Gastroenterología, Barcelona
  - Hospital Vall d'Hebrón Servicio de Aparato Digestivo, Barcelona
  - Hospital General San Jorge de Huesca Servicio de Aparato Digestivo, Huesca
  - Hospital Universitario de Belltvitge Servicio de Cirugía General y Digestiva, L'Hospitalet de Llobregat
  - Hospital Costa del Sol Servicio Digestivo, Marbella
  - Hospital de Ourense Servicio de Aparato Digestivo, Ourense
  - Hospital Universitario de Canarias Servicio de Gastroenterología, Santa Cruz de Tenerife
  - Hospital Clínico Universitario Lozano Blesa Servicio de Aparato Digestivo, Zaragoza
- Yeovil District Hospital NHS Trust Department of Surgery, Yeovil, United Kingdom